CLINICAL TRIAL: NCT03620136
Title: Comparison of Two Techniques of Locoregional Analgesia in Total Knee Prosthesis Surgery : Block to the Adductor Channel Versus Peri-articular Local Infiltrations
Acronym: SALIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 69HCL16_0798; 2016-005213-53 (EudraCT Number)
Record Dates: First submitted 2017-11-14; First posted 2018-08-08 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Analgesic
Keywords: Total knee prosthesis; Adductor canal block; Local peri-articular infiltrations; Postoperative analgesia; Early rehabilitation; Patient Controlled Analgesia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- locoregional analgesia by a block on the adductor channel (Experimental)
  Interventions: Drug: locoregional analgesia by a block on the adductor channel
- locoregional analgesia by periarticular local infiltrations (Experimental)
  Interventions: Drug: locoregional analgesia by periarticular local infiltrations

INTERVENTIONS:
Drug: locoregional analgesia by a block on the adductor channel — The block at the adductor channel will be realized under echo guidance, before the spinal anesthesia, by puncture at the upper 1/3 of the thigh. It will be used echogenic needle adapted to the morphotype of each patient, of varying length from 50mm to 100mm. A single injection of 20mL of ROPIVACAINE 2mg / ml, the efficacy of which should be checked before spinal anesthesia is performed by a cold test.
  Knee analgesia will be supplemented by per-operative infiltration of 50mL of ROPIVACAINE 2mg / ml at the posterior capsule, once the surfaces joints prepared to accommodate the prosthesis and by two placebo infiltrations of 50mL each of physiological saline in the medial and lateral ligaments and in the edges of the incision.
  Arms: locoregional analgesia by a block on the adductor channel
Drug: locoregional analgesia by periarticular local infiltrations — A placebo injection to the adductor channel of 20 mL of physiological serum will be performed in the pre-induction room before surgery, according to the same procedures as the patients of the ACB group.
  During the surgical procedure, patients in the ILA group will receive a total dose of 300mg of ROPIVACAINE 2mg / ml in the form of 3 periarticular injections. The first injection of 50mL of ROPIVACAINE 2mg / ml will be made once the articular surfaces are prepared to receive the prosthesis, at the level of the posterior capsule. The second injection of 50mL of ROPIVACAINE 2mg / ml will be performed once the total knee prosthesis is installed, in the medial and lateral ligaments. Finally, the last injection will also include 50mL of ROPIVACAINE 2mg / ml and will be made in the edges of the incision at the time of closure.
  Arms: locoregional analgesia by periarticular local infiltrations

SUMMARY:
The post-operative pain generated by prosthetic knee replacement surgery is known to be moderate to severe during two or three days following surgery.

The most popular analgesic technique after prosthetic knee replacement surgery remains the femoral block (FB), whether in single injection or continuous infusion. In major knee surgery, FBs provide better analgesia compared to systemic morphine and FBs provide the same analgesia that obtained with epidural analgesia but with fewer associated adverse effects.

Although FBs provide excellent post-operative analgesia after total knee prosthesis, they also provide a significant quadricepsia weakness that increases the risk of severe falls and complications, and hinders the rapid rehabilitation process. For these reasons, alternative analgesic techniques have emerged in recent years.

To avoid the quadricipital motor block generated by FBs, some authors proposed the administration of local anesthetics in the adductor channel, also known as the Hunter channel, in order to produce a pure sensory block. With the development of ultrasound, the adductor channel is easily visualized in the middle of the thigh. This allows the adductor channel block (ACB) to be realized with a high success rate. ACB appears to decrease postoperative pain and morphine consumption. It also significantly improves the ability of patients to walk around after Total Knee Arthroplasty (TKA) surgery.

With the same goal of quadricipital savings, the use of the analgesic technique by periarticular infiltration of local anesthetics (ILA) has spread in recent years, due to the fact that an analgesic technique of simple realization and without apparent danger, and this despite limited evidence of its effectiveness.

The Croix-Rousse Hospital is a university hospital in Lyon with a highly developed orthopedic surgery center, producing approximately 550 TKA per year. During the year 2016, approximately half were benefited from post-operative analgesia management by ACB, and the other half by the implementation of the ILA.

To date few studies have been interested in comparing these two analgesic techniques in knee prosthesis surgery.

ELIGIBILITY:
Inclusion Criteria:

* Major patients (≥18 years),
* Having an American Society of Anesthesiology score (ASA) I to III
* To benefit from first and unilateral prosthetic replacement surgery of knee under spinal anesthesia,
* Having social security scheme,
* Having received informed information and having signed informed consent

Exclusion Criteria:

* Pregnant women (diagnosis of interrogation),
* Breastfeeding women
* Patients under tutorship or curatorship,
* Persons who can not receive sufficient information because of disturbances of superior functions or because of insufficient command of the French language according to the judgment of the investigator,
* A history of chronic neuropathic pain in the leg to be operated on,
* Patients who have undergone prior surgery on the knee to perform surgery,
* Contra-indication to loco-regional anesthesia: known allergy to local anesthetics,
* Contra-indication to the use of ROPIVACAINE: known hypersensitivity to the active substance or other amide-linked local anesthetics, hypovolemia
* A morbid obesity (Body Mass Index (BMI)> 40),
* Severe renal insufficiency (Glomerular Filtration Rate (GFR) <30mL / min),
* Severe hepatic impairment (prothrombin rate PR <50%),
* Heart failure (left ventricular ejection fraction (LVEF)<40%),
* Transplanted patients,
* A history of drug abuse,
* The taking of chronic morphine for 6 months in systematic,
* Any inability to understand visual scale,
* An inability to walk pre-existing,
* Participation in other interventional research, excluding physiological studies and other interventional research that does not interfere with the analysis of the primary endpoint (as determined by the investigator).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-28 (Actual)

PRIMARY OUTCOMES:
the cumulative consumption of MORPHINE | during the first 48 hours following the surgical incision
  cumulative dose of morphine (miligrams). The administration of morphine will be done using a self-controlled analgesic pump (PCA). It will be made available to the patient when he leaves the block. The PCA allows the patient to adapt his consumption of morphine to his needs in analgesics. A nurse regularly reports the amount of morphine that the patient has administered.

SECONDARY OUTCOMES:
Pain at rest | Resting pain will be measured every 4 hours in the first 24 hours, then every 8 hours between 24 and 72 hours
  Postoperative pain will be assessed by a visual scale, graded from 0 to 10, where 0 is a total absence of pain and 10 is the maximum pain. Pain at rest will be measured by the paramedical team
pain in movement | at day 3
  Postoperative pain will be assessed by a visual scale, graded from 0 to 10, where 0 is a total absence of pain and 10 is the maximum pain.
  The movement pain will be assessed daily by the team of physiotherapists for orthostatism, walking, and maximum flexion of the operated knee.
quality of the analgesia offered by the ACB | within 48 hours after the injection to the adductor channel
  the consumption of MORPHINE will be analyzed from different angles in order to evaluate the quality of the analgesia offered by the ACB.
  It will therefore be observed in the ACB group, the time between injection to the adductor channel and the first dose requested on the PCA.
quality of the analgesia offered by the ILA | within 48 hours after the end of surgery
  the consumption of MORPHINE will be analyzed from different angles in order to evaluate the quality of the analgesia offered by the ILA.
  It will be observed the delay between the end of surgery and the use of a first dose of MORPHINE on PCA.
quality of the analgesia | within 48 hours after the surgical incision time
  the curve of consumption of morphine over time from H0 (surgical incision time) to H48 will be established for the 2 arms
Functional capabilities and rehabilitation | at day 3
  The evaluation of the quality and the precocity of the postoperative rehabilitation of the patients will be carried out by the daily measurement of the CAS score (Cumulated Ambulation Score). This score is a validated tool in orthopedic surgery to evaluate daily the recovery of the basic mobility of the patients until return to an autonomy allowing their return home.
Duration of hospitalization | at day 3
  The total duration of hospitalization will be reported after the patient has left, whether it is a return home, or a transfer to a rehabilitation center
Patient satisfaction | at day 3
  overall satisfaction and satisfaction with pain management will be assessed for each patient using a visual scale where 0 is a completely dissatisfied patient and 10 is a fully satisfied patient
Secondary complications due to adductor channel block | Day 0 : At the time of the ACB in the pre-induction room
  All complications related to this gesture should be reported in the case report form : failure (specify the reason), vagal malaise, suspicion of intravenous injection and suspicion of intravascular injection.
Complications secondary to analgesic medications and surgery | at day 3
  Adverse effects associated with the use of MORPHINE, the administration of local anesthetics and related to surgery will be reported in the case report form.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Macabeo, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Croix Rousse Hospital, Lyon, France

REFERENCES:
- [Result] Pic C, Macabeo C, Waissi E, Lasselin P, Raffin M, Pradat P, Lalande L, Lustig S, Aubrun F, Dziadzko M. No Benefit of Adductor Canal Block Compared with Anterior Local Infiltration Analgesia in Primary Total Knee Arthroplasty: A Single-Blinded Randomized Controlled Clinical Trial. J Bone Joint Surg Am. 2023 Feb 1;105(3):231-238. doi: 10.2106/JBJS.22.00745. Epub 2022 Nov 18. PMID 36723467